CLINICAL TRIAL: NCT02090335
Title: Health Promotion and Fitness for Younger and Older Adults With SMI
Acronym: InSHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Stephen J. Bartels, Professor of Psychiatry, of Community and Family Medicine, and of TDI, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Boston In SHAPE; 1R01MH078052 (NIH)
Record Dates: First submitted 2014-03-13; First posted 2014-03-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Schizophrenia; Bipolar Disorder; Schizoaffective Disorder
Keywords: community mental health; health coach; weight loss; fitness; serious mental illness; health promotion
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder; Psychotic Disorders; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- In SHAPE (Experimental): In SHAPE is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Interventions: Behavioral: In SHAPE; Behavioral: Fitness Club Membership
- Fitness Club Membership (Active Comparator): Fitness club membership with education in using the exercise equipment.
  Interventions: Behavioral: Fitness Club Membership

INTERVENTIONS:
Behavioral: In SHAPE — In SHAPE is a health promotion intervention consisting of a fitness club membership and a health promotion coach with basic certification as a fitness trainer, instruction on principles of healthy eating and nutrition, and training in tailoring individual wellness plans to the needs of persons with serious mental illness.
  Arms: In SHAPE
Behavioral: Fitness Club Membership — Fitness club membership with education in using the exercise equipment.

SUMMARY:
The goal of this project, which has not changed, is to improve the health and fitness of persons with serious mental illness (SMI) using an innovative model: In SHAPE Lifestyles. Participants are randomly assigned to the In SHAPE program or Health Club Membership and Education only.

The three specific aims of this study are to:

1. To compare the treatment groups with respect to improvement in physical fitness outcomes, including: (a) health behaviors (engagement in exercise and diet changes); and (b) indicators of physical fitness.
2. To compare the treatment groups with respect to improvements in mental health outcomes, including negative symptoms, depression, and self-efficacy.
3. To explore differences in the treatment groups with respect to psychosocial functioning, health status, and acute service use, and the effects of selected demographic, clinical, and health behavior variables on primary outcomes.

DETAILED DESCRIPTION:
Individuals with SMI die 10-25 years earlier than the general population and have disproportionately greater rates of medical comorbidity and disability associated with high rates of obesity, sedentary lifestyle, metabolic syndrome, and poor dietary habits. Despite greater costs and adverse outcomes associated with the combination of mental illness and poor physical health, little attention has been paid to the development of health promotion interventions designed to address the needs of the high-risk group of people with SMI. This study is testing an innovative approach to reducing these problems and developing a program that will potentially have a downstream effect on early mortality for the vulnerable population of people with SMI.

ELIGIBILITY:
Inclusion Criteria:

* age 21 or older
* serious mental illness defined by an axis I diagnosis of major depression, bipolar disorder, schizoaffective disorder, or schizophrenia
* persistent impairment in multiple areas of functioning (e.g., work, school, self-care)
* body mass index (BMI) greater than 25
* able and willing to provide informed consent
* on stable pharmacological treatment (same psychiatric medications over prior 2 months)

Exclusion Criteria:

* residing in nursing home or other institution
* diagnosis of dementia or significant cognitive impairment (MMSE<24)
* unable to walk one city block
* pregnant or planning to become pregnant within the next 18 months
* unable to speak English
* terminal illness with life expectancy<1 year
* current diagnosis of an active substance dependence disorder

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2007-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 3-, 6-, 9-, 12-, and 18-months
  Change in weight over time was measured at baseline, 3-, 6-, 9-, 12-, and 18-months. Measures were weight (kg) and body mass index (kg/m2).

SECONDARY OUTCOMES:
Change in Dietary Behaviors | Baseline, 6-, 12-, and 18-months
  Change in dietary behaviors was assessed over time using a scale adapted from the Stages of Change Modified Motivational Interviewing instrument focused on dietary behaviors and physical activity.
Change in Dietary Intake | Baseline, 6-, 12-, and 18-months
  Change in dietary intake over time was assessed using the Brief Block Food Frequency Questionnaire and nutrient analysis was conducted with NutritionQuest using a nutrient database developed from the USDA Nutrient Database for Standard Reference.
Change in Serum lipids | Baseline, 6-, 12-, and 18-months
  Change in serum lipids over time was measured using the CardioChek PA Analyzer, a hand-held dual testing system that produces values for total cholesterol, LDL, HDL, and triglycerides using a multi-panel test strip and a single drop of blood acquired with a finger prick.
Change in Blood Pressure | Baseline, 6-, 12-, and 18-months
  Change in systolic and diastolic blood pressure over time was measured using a blood pressure cuff.
Change in Cardiorespiratory Fitness | Baseline, 6-, 12-, and 18-months
  Change in cardiorespiratory fitness over time was measured using the 6 Minute Walk Test (distance in m that a participant can walk in 6 minutes).
Change in Physical Activity | Baseline, 3-, 6-, 9-, 12-, and 18-months
  Change in self-reported physical activity was measured over time using the short-form International Physical Activity Questionnaire (IPAQ).

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Bartels, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (3):
- United States (3):
  - Baycove Human Services, Boston, Massachusetts
  - Massachusetts Mental Health Center, Boston, Massachusetts
  - Vinfen, Cambridge, Massachusetts

REFERENCES:
- [Derived] Naslund JA, Aschbrenner KA, Pratt SI, Lohman MC, Scherer EA, McHugo GJ, Marsch LA, Unutzer J, Bartels SJ. Association Between Cardiovascular Risk and Depressive Symptoms Among People With Serious Mental Illness. J Nerv Ment Dis. 2017 Aug;205(8):634-640. doi: 10.1097/NMD.0000000000000669. PMID 28240625
- [Derived] Bartels SJ, Pratt SI, Aschbrenner KA, Barre LK, Naslund JA, Wolfe R, Xie H, McHugo GJ, Jimenez DE, Jue K, Feldman J, Bird BL. Pragmatic replication trial of health promotion coaching for obesity in serious mental illness and maintenance of outcomes. Am J Psychiatry. 2015 Apr;172(4):344-52. doi: 10.1176/appi.ajp.2014.14030357. Epub 2014 Dec 12. PMID 25827032